CLINICAL TRIAL: NCT01698242
Title: Reduction in Hospitalizations in Low-Income Patients With Heart Failure
Brief Title: The Congestive Heart Failure Adherence Redesign Trial
Acronym: CHART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lynda Powell, PhD, MEd (Other)
Collaborators: Cook County Health (Other Government); Sinai Health System (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor-Investigator, Lynda Powell, PhD, MEd, Principal Investigator, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10030801
Record Dates: First submitted 2012-06-12; First posted 2012-10-02 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure, Congestive; Cardiovascular Diseases; Heart Diseases
Keywords: Heart failure; Self-Management; Behavioral Clinical Trial
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Training (Experimental): The Enhanced Training intervention follows a multi-level strategy in which both the patient and their PCP are intervened upon concurrently. Randomization occurs at the PCP-level, that is, patients are assigned to the Enhanced Training group only if their PCP has been enrolled and randomized to this group. Descriptions of the intervention on the PCP-level and patient-level are provided in the intervention section.
  Interventions: Behavioral: Enhanced Training
- Enhanced Education (Active Comparator): The Enhanced Education intervention follows a multi-level strategy in which both the patient and their PCP are intervened upon concurrently. The intervention strategy revolves around providing nominal information through the mail. Randomization occurs at the PCP-level; that is, patients are assigned to the Enhanced Education group only if their PCP already has been enrolled and randomized to this group. Description of the intervention on the PCP-level and patient-level is provided in the intervention section.
  Interventions: Behavioral: Enhanced Education

INTERVENTIONS:
Behavioral: Enhanced Training — PCP-Level: A PCP randomized to the Enhanced Training (ET) group will receive: 1) a full and pocket sized copy of the current AHA Heart Failure (HF) Guidelines; 2) a summary of their patient's data collected at baseline, 6-month, and 30-month in-person study visits; and 3) an invitation to complete the CHART-designed online course in HF management for CME credit.
  Patient Level: The ET patient-level intervention uses Community Health Workers (CHWs) to assist the patient in learning self-management behaviors to reduce the risk of hospitalization. The key objectives are to: improve heart failure knowledge; encourage use of HF management tools; and facilitate development of self-management skills. Each participant receives at least: six AHA educational mailings, six monthly home visits, and 18 phone calls by CHWs within the first six months of the intervention. The CHW then conducts monthly telephone visits for the subsequent two years (for a total of 30 months of follow-up).
  Arms: Enhanced Training
Behavioral: Enhanced Education — The Enhanced Education (EE) intervention follows a multi-level strategy in which both the patient and their PCP are intervened upon concurrently. The intervention provides nominal information through the mail. Randomization occurs at the PCP-level; patients are assigned to the EE group only if their PCP already has been randomized to this group.
  PCP Level: Upon randomization to the EE group each PCP will receive a full-sized copy of the current American Heart Association (AHA) Heart Failure Guidelines within thirty days after randomization.
  Patient Level: Upon their assignment to the EE group, patients will receive: Six AHA Tip-Sheet mailings (one Tip-Sheet to be mailed each of the first six months following group assignment); a telephone call, made by the CHART Research Assistant (RA), completed once during each of the first six months following group assignment and only to confirm that the patient received the Tip-Sheet mailing for that month.
  Arms: Enhanced Education

SUMMARY:
The purpose of this study is to test whether a culturally sensitive self-management (SM) intervention, compared to an education only control, will reduce all-cause hospital days in patients with mild to moderate heart failure and household income less than $30,000 per year.

DETAILED DESCRIPTION:
The purpose of the CHART research study is to assess the value of a novel multi-level intervention for low-income patients recently hospitalized with heart failure relative to providing education alone (both strategies are described in detail in the Intervention section below). The investigators refer to their novel intervention strategy as 'Enhanced Training' and their education-only strategy the investigators refer to as 'Enhanced Education'. These two strategies of participant follow-up will be assessed and compared by analyzing patient's all-cause hospital days over a 2.5-year follow-up period (the investigators note that, for patients with heart failure, the average number of such all-cause hospital days over a 2.5-year period has tripled over the past 25 years). The Enhanced Training strategy aims to improve patient receipt of evidence-based therapy by: 1) activating patients using a culturally sensitive approach that might better resonate with the investigators predominantly urban, African-American and Hispanic, target population; 2) providing timely and useful information to the primary care provider; and 3) promoting effective communication between patients and their primary care provider. The Enhanced Education strategy is less intrusive and aims to provide patients and primary care providers with appropriate educational materials via mail. The primary aims of this research study are to determine if Enhanced Training and/or Enhanced Education will improve: patient adherence to drug therapy and salt restriction, health care provider adherence to evidence-based guidelines, and patient functional capacity and quality of life. Secondary aims will include assessing impact of the interventions on CRP and BNP, which are two key biomarkers of heart failure progression.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (PCP) 1. Provider must be the health professional who is managing the potential patient enrollee's heart failure medication(s).

Inclusion Criteria (Patients)

1. Participant has been diagnosed with Heart Failure (HF),
2. Self reported family income is less than $30,000/year,
3. Has experienced at least one hospitalization for acute, decompensated, HF within the previous 6 months based upon:

   1. Being admitted for symptoms of HF (ex: peripheral edema, shortness of breath and fatigue), and
   2. responding to anti-failure therapy such as diuretics and other anti-failure therapy such as ACE Inhibitors, ARBs, or Beta blockers.
4. Has evidence of systolic dysfunction, defined by an ejection <50 by 1 of 3 methods: echocardiography, radiographic contrast ventriculography, or nuclear ventriculography; done within the last year.
5. Age ≥ 18 years
6. Currently resides in Cook County, Illinois.
7. Speaks English or Spanish.
8. The primary care provider (PCP) has consented and has no more than 12 patients enrolled.
9. Completed the informed consent process.
10. Successfully completed the 30-day run-in period and study baseline visit

Exclusion Criteria:

Exclusion Criteria (PCP)

Health providers will be excluded from enrollment if they are:

1. Still in their residency or training period,
2. A member of the CHART research staff.

Exclusion Criteria (Patients)

Patients will be excluded from enrollment if they have:

1. An uncertain 12-month prognosis.

1. Listed for imminent cardiac transplant.
2. Has an advanced directive of "Do not resuscitate".
3. Has uncertain 12-Month Prognosis, as adjudicated by the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total number of all cause hospitalization days | Measured over the 30 month patient participant follow-up period
  Participant's are queried quarterly concerning any hospitalizations occuring since the previous contact. These self-reported events are then confirmed via study adjudication of pertinent acquired hospital medical records. Analysis of the primary outcome will consist of comparing mean total number of all-cause hospitalization days between the two intervention groups. Analyses will also be performed with respect to the following pre-determined subgroups: (Primary Healthcare Provider subgroups) medical specialty, academic rank, "adherent" to evidence-based guidelines at baseline, and number of years since certification; (Patient Participant subgroups) age, gender, ethnicity, insurance status, years of education, health literacy, number of comorbidities, medication adherence at baseline, heart failure functional capacity, baseline BNP, presence of major stress and/or psychological trauma, perceived social support, number of years since first heart failure diagnosis, and self-efficacy

SECONDARY OUTCOMES:
Total number of heart failure related hospitalization days | measured over the 30 month patient participant follow-up period
  Participants are queried quarterly during the 30-month study follow-up period as to any hospitalizations that occurred since the previous study contact. These self-reported events are then determined to be heart failure related via study adjudication of pertinent acquired hospital medical records.
Health Care Costs | Measured over the 30 monthstudy follow-up period
  Participant's are queried quarterly during study follow-up as to any hospitalizations, nursing home stays, or home health care episodes since the previous study contact. The costs of these self-reported events are then determined via study adjudication of collected hospital medical record. (costs of emergency room visits will be considered separately).
Distance traveled during th Six-Minute Walk test | This test is administered during in-person participant assessment visits conducted at baseline and at 6 and 30 months following treatment assignmentMeasured over/after 30 months
  The Six-Minute Walk test is a supervised patient performance measure used in heart failure assessment. Standard six-minute walk safety procedures are used to ensure participant safety during conduct of this test.
The Kansas City Cardiomyopathy Questionnaire | This questionnaire is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  This questionnaire is a 23-item, self-administered questionnaire that quantifies physical function, symptoms, social function, self-efficacy, and quality of life for patients with heart failure. Scores range from 0 to 100 where higher scores indicate better function.
Patient Medication Adherence | Adherence is measured at baseline and at 6 and 30 months following treatment assignment
  Medication adherence will be assessed by tracking a single heart failure medication (an ACE, ARB, Beta-Blocker, or diuretic typically). Tracking will be done using a MEMS™ electronic pill monitoring cap from AARDEX and comparing the medication regimen observed to the regimen prescribed by their health care provider. To ensure participant safety, we have instituted a study protocol to help ensure participants' routine medication-taking behavior is not compromised by the use of an electronic pill cap device.
CALS Food Frequency Questionnaire (Salt Intake) | This questionnaire is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  To determine salt intake over the past week, the CALS Food Frequency Questionnaire will be used. This questionnaire has been specially developed to focus on dietary items that are main sources of sodium. It is computer-scored and provides data on total sodium consumed and can track changes in sodium intake over time.
Self-Efficacy of Heart Failure Self-Management | This is a questionnaire that is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  The Self-Efficacy at Self-Management Scale directly assesses confidence in the use of the 5 specific self-management skills that are a target of the Enhanced Training intervention.
EQ-5D Visual Analog Scale (VAS) with Time Trade-Off (TTO) Utility Score | This is a questionnaire that is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  The EQ-5D self-report questionnaire consists of a 5-item health state assessment (rated as 1=none, 2=some, 3=severe), to produce an index score. Responses to the health state items can be converted to a time trade-off (TTO) utility score, where 1 represents perfect health and 0 represents death (negative utilities are possible, representing states worse than death). A visual analog scale (VAS) can be applied, scored from 0 to 100, where higher scores are better. EQ-5D index score can be used to produce health utilities and to estimate quality-adjusted life-years (QALYs) gained or lost.
Biomarkers of heart failure progression | Assessed during in-person participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  Two biomarkers are accessed via blood assays; High sensitivity C-reactive protein (hsCRP) and B-type natriuretic peptide (BNP). Plasma hs CRP, an inflammatory marker, is associated with worse heart failure outcomes. Heart failure treatment reduces hsCRP. B-type natriuretic peptide (BNP) is a biomarker of myocyte stress. Standard safety procedures are used in performing the participant blood draw required for this measure.
PHQ9 (Depression) | This is a questionnaire that is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  The PHQ9 is comprised of 9 self-reported items answered in "Not at all = 0; Several days = 1; More than half the days = 2; Nearly every day = 3" format summed to yield score between 0-27. Higher score indicates more severe depression symptoms.
Past Stressor Events | This is a questionnaire that is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  : This 10-item questionnaire assesses a list of major stressful life events, focusing on several important domains: severe illness, death of a loved one, family conflict/divorce, financial problems, and exposure to neighborhood or workplace violence, including sexual abuse and rape, assessed as Yes/No/Refusal responses.
Traumatic Stress Survey (Composite International Diagnostic Interview) | This survey that is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  A 11-item questionnaire assesses a list of Traumatic Stress life events , including: Being in a natural disaster, a serious accident, being attacked with or without a weapon, military combat or in a war zone, sexual abuse and rape, and other situations extraordinarily stressful situations. Responses are Yes/No/Don't Know/Refusal. If a participant indicates an event occurred the frequency is assessed with 4 possible responses from never=0, 1 time=1, 2-3 times =3, and 4 or more times = 4.
PCL-Civilian Short Form | This is a questionnaire that is administered during participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  This 6-item screen for post-traumatic stress disorder (PTSD) was derived empirically from the PCL-C Questionnaire for use in primary care settings. It contains 2 items from each of 3 subscales that correlated most highly with the overall subscale score. The 3 subscales are: Re-Experiencing, Avoidance, and Hyper-Arousal. Respondents rate items on a 5-point scale (ranging from 1 = "Not at all" to 5 = "Extremely"). The short scale has been found to have good reliability and validity and is used as an indication of symptoms of PTSD.
Modified Global Adherence Indicator (mGAI3) | This is assessed at baseline and at 6 and 30 months following participant treatment assignment.
  This physician adherence indicator is based on prescribing the three pharmacological classes of HF medications (ACEI/ARB, beta-blockers, and aldosterone antagonists). This endpoint is assessed by reviewing the most recent pertinent outpatient medical record at each time point for each participant. The modified Global Adherence indicator (mGAI) is computed for each participant by calculating the proportion of indicated care (across three therapeutic classes). The higher mGAI indicates better adherence.
PCP Adherence to blood pressure goal | Patient participant blood pressure is assessed during in-person participant assessments conducted at baseline and at 6 and 30 months following treatment assignment.
  For each enrolled PCP, the proportion of their patients participating in the study achieving blood pressure below 130/80 mm Hg during study assessments is computed.
Total number of heart failure hospitalizations and emergency room visits. | Measured over the 30 month patient participant follow-up period.
  Total number of heart failure hospitalizations and heart failure emergency room visits, separately and combined, overall and by subgroups indicated above.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda H. Powell, PhD, Principal Investigator — Chairperson and Professor
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Calvin JE, Shanbhag S, Avery E, Kane J, Richardson D, Powell L. Adherence to evidence-based guidelines for heart failure in physicians and their patients: lessons from the Heart Failure Adherence Retention Trial (HART). Congest Heart Fail. 2012 Mar-Apr;18(2):73-8. doi: 10.1111/j.1751-7133.2011.00263.x. Epub 2011 Nov 3. PMID 22432552
- [Background] Powell LH, Calvin JE Jr, Mendes de Leon CF, Richardson D, Grady KL, Flynn KJ, Rucker-Whitaker CS, Janssen I, Kravitz G, Eaton C; Heart Failure Adherence and Retention Trial Investigators. The Heart Failure Adherence and Retention Trial (HART): design and rationale. Am Heart J. 2008 Sep;156(3):452-60. doi: 10.1016/j.ahj.2008.05.011. PMID 18760125
- [Background] de Leon CF, Grady KL, Eaton C, Rucker-Whitaker C, Janssen I, Calvin J, Powell LH. Quality of life in a diverse population of patients with heart failure: BASELINE FINDINGS FROM THE HEART FAILURE ADHERENCE AND RETENTION TRIAL (HART). J Cardiopulm Rehabil Prev. 2009 May-Jun;29(3):171-8. doi: 10.1097/HCR.0b013e31819a0266. PMID 19471136
- [Background] Powell LH, Calvin JE Jr, Richardson D, Janssen I, Mendes de Leon CF, Flynn KJ, Grady KL, Rucker-Whitaker CS, Eaton C, Avery E; HART Investigators. Self-management counseling in patients with heart failure: the heart failure adherence and retention randomized behavioral trial. JAMA. 2010 Sep 22;304(12):1331-8. doi: 10.1001/jama.2010.1362. PMID 20858878
- [Background] Rucker-Whitaker C, Flynn KJ, Kravitz G, Eaton C, Calvin JE, Powell LH. Understanding African-American participation in a behavioral intervention: results from focus groups. Contemp Clin Trials. 2006 Jun;27(3):274-86. doi: 10.1016/j.cct.2005.11.006. Epub 2006 Jan 19. PMID 16427365